CLINICAL TRIAL: NCT06230939
Title: Examination of Factors Associated With Fatigue in Individuals Diagnosed With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Asli Demirtaş, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: Gazi University-05.09.2023.3
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Fatigue
Keywords: Parkinson's disease; Fatigue; Examination
MeSH Terms: conditions — Parkinson Disease; Fatigue | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's Disease Group: The study will be conducted in collaboration with Gazi University Faculty of Health Sciences and Nigde Omer Halisdemir University. The study data will be obtained from individuals diagnosed with PD admitted to the Neurology Outpatient Clinic of Nigde Omer Halisdemir University Training and Research Hospital. Necessary permissions were obtained from all institutions. All evaluations will be collected in a single meeting using the face-to-face interview method. It is calculated that 80% power will be reached with a margin of error of 0.05 when 84 individuals diagnosed with PD are included in the study.
  Interventions: Other: Examination

INTERVENTIONS:
Other: Examination — Individual characteristics of the patients (gender, age, height, body weight, marital status, education level, dominant extremity, smoking and alcohol consumption habits, use and type of assistive device, how many years the assistive device has been used) and disease-related (year of diagnosis, disease duration Information (such as CV, family history, medications used, surgeries) will be questioned. HYE and UPDRS will be used for disease staging and grading. PFS-16 will be used to evaluate fatigue and MMSE will be used to evaluate sleep. In addition, "Timed Up and Go (TUG)" will be applied for lower extremity performance evaluation. All evaluations will be collected in a single meeting using the face-to-face interview method.

SUMMARY:
Fatigue is defined as an overwhelming feeling of weariness, lack of energy, and a feeling of exhaustion. It is common in Parkinson's Disease (PD) and is one of the most disabling symptoms. Fatigue is affected by motor and non-motor symptoms in individuals diagnosed with PD. As a result of this impact, it manifests itself as difficulty in initiating and continuing mental and physical tasks. This study aims to examine the fatigue of individuals diagnosed with PD and the factors associated with this fatigue.

DETAILED DESCRIPTION:
The study will be carried out in cooperation with Gazi University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation and Nigde Omer Halisdemir University, and the study data will be collected from individuals diagnosed with PD who applied to the Neurology Polyclinic of Nigde Omer Halisdemir University Training and Research Hospital. Necessary permissions have been obtained from all institutions. Modified Hoehn&Yahr staging (HYS) and Unified Parkinson's Disease Rating Scale (UPDRS and its subtests) will be used for disease staging and grading. Parkinson's Fatigue Scale-16 (PFS-16) to evaluate fatigue, Parkinson's Disease Sleep Scale-2 (PDSS-2) to evaluate sleep, Hospital Anxiety and Depression Scale (HAD) to evaluate depression and anxiety, Mini-Mental to evaluate cognitive status (MMSE) will be used. In addition, "Timed Up and Go (TUG)" will be applied for lower extremity performance evaluation. All evaluations will be collected in a single meeting using the face-to-face interview method. It is calculated that 80% power will be reached with a margin of error of 0.05 when 84 individuals diagnosed with PD are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Being diagnosed with PD by a neurologist,
* Having stable medical treatment,
* Being able to stand independently for at least 60 seconds without any assistive device,
* Having received 18 points or more according to the MMSD evaluation.

Exclusion Criteria:

* Being illiterate or unable to communicate in Turkish,
* Having undergone a surgery that may affect lower extremity functions,
* Diabetes mellitus is a diagnosis of another neurological and rheumatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research will be carried out in cooperation with Gazi University Faculty of Health Sciences and Nigde Omer Halisdemir University. Study data will be obtained from individuals diagnosed with PD who apply to Nigde Omer Halisdemir University Training and Research Hospital Neurology Polyclinic. Necessary permissions were obtained from all institutions.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Parkinson Fatigue Scale-16 (PFS-16); | Baseline
  PFS-16, consists of 16 items designed to evaluate the impact of fatigue on daily life and its physical dimensions. The scale allows measuring the presence of fatigue (7 items) and its impact on daily function (9 items). Individuals are asked to respond to statements about fatigue on a 5-point Likert scale between 1 (strongly disagree) and 5 (strongly agree).
Hospital Anxiety and Depression Survey (HAD) | Baseline
  Each item of the scale, which consists of 14 items, is scored between 0 and 3. For anxiety and depression values, 0-7 points are considered normal, 8-10 points are considered borderline, and 11 points and above are considered abnormal. The validity and reliability of this scale in Turkish has been established.
Parkinson's Disease Sleep Scale-2 (PDSS-2) | Baseline
  The scale is a 5-point Likert type (4: Very often, 6-7 days a week; 3: Frequently, 4-5 days a week; 2: Sometimes, 2-3 days a week; 1: Occasionally, 1 day a week; 0: Never) consists of 15 items. The scale includes general night sleep quality (item 1), falling asleep (item 2), insomnia (item 3), night restlessness (items 4 and 5), night psychosis (items 6 and 7), nocturia (item 8). . and items 9), night motor symptoms (items 10, 11, 12 and 13), waking up rested (item 14) and sleep-disordered breathing (item 15) are evaluated.
Time Up and Go Test (TUG) | Baseline
  Timed get up and go test is used for functional evaluation of patients. This test is important in terms of evaluating patients' walking speed as well as testing their ability to maintain balance. In the test application, after the patient gets up from the chair without back support, he walks three meters to the marked area, turns back, and on the way back, the time to sit on the chair is calculated by walking three meters again. The test is repeated three times and the average in seconds is recorded.

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | Baseline
  MMSE will be used to evaluate cognitive functions. The mini mental test is categorized under five main headings. It consists of 11 items including orientation (10 points), recording memory (3 points), attention and calculation (5 points), recall (3 points) and language (9 points). It is evaluated over 30 points in total. A score between 24-30 points is defined as normal, 18-23 points as mild dementia, and 17 points and below as severe dementia. The average administration time of the test is 10 minutes. Patients scoring 18 and above will be included in the study.
Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline
  Unified Parkinson's Disease Rating Scale (UPDRS) is a scale created to evaluate the motor performance, mental and spiritual status, and daily life activities of patients diagnosed with PD. The scale consists of a total of 4 sections and 42 items. In the first part, non-motor symptoms such as thoughts, behavior and affect; In the second part, activities of daily living; motor symptoms in the third part; In the fourth section, treatment complications are evaluated. Each item is scored between 0 (no symptoms or signs) and 4 (the most severe symptom or sign possible).
Modified Hoehn-Yahr Evaluation (MHYE) | Baseline
  Modified Hoehn-Yahr Evaluation (MHYE) used to define the disease stage of patients diagnosed with PD. According to MHYE, the disease consists of 8 stages. It is stated that the disease symptoms worsen as the stage progresses.
Interview Form | Baseline
  All evaluations will be carried out by face-to-face interview method. Individual characteristics of the patients (gender, age, height, body weight, marital status, education level, dominant extremity, smoking and alcohol consumption habits, use and type of assistive device, how many years the assistive device has been used) and disease-related (year of diagnosis, disease duration Information (such as CV, family history, medications used, surgeries) will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: İlke KESER, Prof. Dr., Study Director — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Ankara
  - Nigde Omer Halisdemir University, Niğde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Opara J, Malecki A, Malecka E, Socha T. Motor assessment in Parkinson;s disease. Ann Agric Environ Med. 2017 Sep 21;24(3):411-415. doi: 10.5604/12321966.1232774. Epub 2017 May 11. PMID 28954481
- [Background] Ascherio A, Schwarzschild MA. The epidemiology of Parkinson's disease: risk factors and prevention. Lancet Neurol. 2016 Nov;15(12):1257-1272. doi: 10.1016/S1474-4422(16)30230-7. Epub 2016 Oct 11. PMID 27751556